CLINICAL TRIAL: NCT01304316
Title: Cardiovascular Changes and Tetracaine Pharmacokinetics Following Intranasal Administration of Standard and High Doses of Kovacaine Mist (Tetracaine Hydrochloride With Oxymetazoline Hydrochloride) in Healthy Volunteers
Brief Title: Dose-Escalation Safety and Pharmacokinetic Study of K305
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Renatus, LLC (Industry)
Collaborators: Ground Zero Pharmaceuticals (Industry); Rho, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SR 2-02
Record Dates: First submitted 2011-02-18; First posted 2011-02-25 (Estimated); Results first posted 2017-08-31 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2017-07

CONDITIONS: Anesthesia
MeSH Terms: interventions — Tetracaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Kovacaine Nasal Spray (Experimental): Tetracaine HCl 3% and Oxymetazoline HCl 0.05%: 6 sprays of 0.1 mL - total of 18 mg tetracaine HCl and 0.3 mg oxymetazoline HCl followed by 12 sprays of 0.1 mL - total of 36 mg tetracaine HCl and 0.6 mg oxymetazoline HCl
  Interventions: Drug: Tetracaine HCl 3% and Oxymetazoline HCl 0.05%

INTERVENTIONS:
Drug: Tetracaine HCl 3% and Oxymetazoline HCl 0.05% — Tetracaine HCl 3% and Oxymetazoline HCl 0.05%
  Other Names: Kovacaine Nasal Spray

SUMMARY:
The purpose of this study is to determine the pharmacokinetics/pharmacodynamics and safety of a nasal spray containing the anesthetic drug tetracaine in combination with oxymetazoline

DETAILED DESCRIPTION:
The purpose of this study was to determine the safety and pharmacokinetics of the standard dose of intranasal Kovacaine Mist of 0.6 mL (18 mg tetracaine HCl with 0.3 mg oxymetazoline HCl) and a proposed maximum recommended dental dose of 1.2 mL (36 mg tetracaine HCl with 0.6 mg oxymetazoline HCl). The primary objectives were to determine if either dose significantly changed blood pressure readings (systolic and diastolic), pulse rate, or oxygen saturation levels from baseline pretreatment values and to determine the safety profile of both doses. The secondary objectives were to establish the pharmacokinetics of oxymetazoline, tetracaine, and its major metabolite (parabutylaminobenzoic acid) following the intranasal administration of both doses. Each subject received the standard dose (3 sprays in each nostril with 4 minutes between each pair of sprays) followed 1 to 3 weeks later by the high dose (as 6 sprays in each nostril).

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 65 years of age
* BMI between19 and 29 kg/m2
* Sufficiently healthy as determined by the investigator to receive the test medications and undergo the scheduled study procedure
* Can breathe through both nostrils
* Females of child-bearing potential must have a negative urine pregnancy test and must have been using adequate means of birth control for at least one month prior to study entry and during the study
* Screening BP ≤ 140/90
* Screening SpO2 ≥ 96
* Can understand and sign the informed consent document
* Can communicate with the investigator
* Can understand and comply with the requirements of the protocol.

Exclusion Criteria:

* A clinically relevant history or presence of respiratory, thyroid, gastrointestinal, renal, hepatic, hematological, lymphatic, cardiovascular, psychiatric, neurologic, musculoskeletal, genitourinary, infective, inflammatory, immunological, dermatological, or connective tissue disease or disorder or a clinically relevant history or presence of narrow angle glaucoma and in men benign prostatic hypertrophy, Hashimoto"s Thyroiditis, lymphocytic thyroiditis, or uncontrolled diabetes
* Clinically significant abnormalities in laboratory values
* Clinically relevant sinus/nasal surgical history
* Current condition, such as nasal congestion or sinus infection, that may influence responses to study medication
* History of recurrent nose bleeds
* History of pseudocholinesterase deficiency or previous prolonged paralysis with succinylcholine or "difficulty waking up from general anesthesia"
* Allergic to or intolerant of tetracaine, benzocaine, other ester local anesthetics, or para-aminobenzoic acid (as found in PABA-containing sunscreens)
* Allergic to or intolerant of oxymetazoline or preservatives found in these solutions
* History of alcoholism and/or drug abuse
* Have taken a monamine oxidase inhibitor, or vasopressor drug within the past 3 weeks
* Have received or taken local anesthetics within 72 hours of the first or second treatment visits
* Are nursing, pregnant, suspected of being pregnant, or trying to become pregnant (Females will be required to take a urine pregnancy test at each study visit to rule out pregnancy)
* Have used any investigational drug and/or participated in any clinical trial within 30 days of baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-09; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elliot V Hersh, DMD, MS, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, School of Dental Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Kovacaine Nasal Spray
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Kovacaine Nasal Spray
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.2 (7.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Cmax of Oxymetazoline
Description: Extra-vascular, non-compartmental analysis is used to derive pharmacokinetic parameters; estimated from observed plasma concentration values, the dose administered, the AUCs, and the terminal elimination phase rate constant for each dose group
Time Frame: Baseline, 5, 10, 15, 20, 25, 30, 40, 50, 60, 70, 80, 90, 100, 110, 120 minutes
Population: Only 11 subjects in the 0.3 mg dose group had sufficient concentration levels to calculate Cmax.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Kovacaine Nasal Spray
Number analyzed (Participants) | 12
ng/mL
  0.3 mg: number analyzed (Participants) | 11
  0.3 mg | 1.45 (0.473)
  0.6 mg | 2.05 (0.748)

2. Primary Outcome: Cmax of Tetracaine
Description: as for outcome 1
Time Frame: Baseline, 5, 10, 15, 20, 25, 30, 40, 50, 60, 70, 80, 90, 100, 110, 120 minutes
Population: Only 4 subjects in the 18 mg dose group and 7 subjects in the 36 mg dose group had sufficient concentration levels to calculate Cmax.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Kovacaine Nasal Spray
Number analyzed (Participants) | 12
ng/mL
  18 mg: number analyzed (Participants) | 4
  18 mg | 0.243 (0.113)
  36 mg: number analyzed (Participants) | 7
  36 mg | 1.15 (2.45)

3. Primary Outcome: Cmax of PBBA
Description: as for outcome 1
Time Frame: Baseline, 5, 10, 15, 20, 25, 30, 40, 50, 60, 70, 80, 90, 100, 110, 120 minutes
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Kovacaine Nasal Spray
Number analyzed (Participants) | 12
ng/mL
  Standard Dose | 492 (189)
  High Dose | 886 (289)

4. Primary Outcome: Half Life of Oxymetazoline
Description: as for outcome 1
Time Frame: Baseline, 5, 10, 15, 20, 25, 30, 40, 50, 60, 70, 80, 90, 100, 110, 120 minutes
Population: Only 7 subjects in the 0.3 mg dose group and 0.6 mg dose group had sufficient concentration levels to calculate the half life.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Kovacaine Nasal Spray
Number analyzed (Participants) | 12
h
  0.3 mg: number analyzed (Participants) | 7
  0.3 mg | 2.32 (0.86)
  0.6 mg: number analyzed (Participants) | 7
  0.6 mg | 1.72 (0.46)

5. Primary Outcome: Half Life of Tetracaine
Description: as for outcome 1
Time Frame: Baseline, 5, 10, 15, 20, 25, 30, 40, 50, 60, 70, 80, 90, 100, 110, 120 minutes
Population: An insufficient number of tetracaine plasma concentrations existed in each subject to determine a half life for tetracaine
Arm/Group | Kovacaine Nasal Spray
Number analyzed (Participants) | 0

6. Primary Outcome: Half Life of PBBA
Description: as for outcome 1
Time Frame: Baseline, 5, 10, 15, 20, 25, 30, 40, 50, 60, 70, 80, 90, 100, 110, 120 minutes
Population: Only 8 subjects in the standard dose group and 11 subjects in the high dose group had sufficient concentration levels to calculate Cmax.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Kovacaine Nasal Spray
Number analyzed (Participants) | 12
h
  Standard dose: number analyzed (Participants) | 8
  Standard dose | 1.00 (0.33)
  High dose: number analyzed (Participants) | 11
  High dose | 1.01 (0.32)

7. Secondary Outcome: Pulse Oximetry Maximum Change From Baseline
Time Frame: Baseline, 5, 10, 15, 20, 25, 30, 40, 50, 60, 70, 80, 90, 100, 110, 120 minutes
Measure: Mean (Standard Deviation); unit: % oxygen
Arm/Group | Kovacaine Nasal Spray
Number analyzed (Participants) | 12
% oxygen
  Standard K305 Dose | 0.9 (0.9)
  High K305 Dose | 0.3 (0.65)

8. Secondary Outcome: Diastolic BP Maximum Change From Baseline
Time Frame: Baseline, 5, 10, 15, 20, 25, 30, 40, 50, 60, 70, 80, 90, 100, 110, 120 minutes
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Kovacaine Nasal Spray
Number analyzed (Participants) | 12
mmHg
  Standard K305 Dose | 10.8 (7.74)
  High K305 Dose | 11.7 (8.28)

9. Secondary Outcome: Systolic BP Maximum Change From Baseline
Time Frame: Baseline, 5, 10, 15, 20, 25, 30, 40, 50, 60, 70, 80, 90, 100, 110, 120 minutes
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Kovacaine Nasal Spray
Number analyzed (Participants) | 12
mmHg
  Standard K305 Dose | 10.7 (7.67)
  High K305 Dose | 14.7 (8.60)

10. Secondary Outcome: Pulse Rate Maximum Change From Baseline
Time Frame: Baseline, 5, 10, 15, 20, 25, 30, 40, 50, 60, 70, 80, 90, 100, 110, 120 minutes
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Kovacaine Nasal Spray
Number analyzed (Participants) | 12
bpm
  Standard K305 Dose | 5.2 (4.39)
  High K305 Dose | 8.5 (8.25)

ADVERSE EVENTS:
Time Frame: 2 to 3 weeks
Groups:
- Standard K305 Dose: Tetracaine HCl 3% and Oxymetazoline HCl 0.05%: 6 sprays of 0.1 mL - total of 18 mg tetracaine HCl and 0.3 mg oxymetazoline HCl
- High K305 Dose: Tetracaine HCl 3% and Oxymetazoline HCl 0.05%: 12 sprays of 0.1 mL - total of 36 mg tetracaine HCl and 0.6 mg oxymetazoline HCl
Arm/Group | Standard K305 Dose | High K305 Dose
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 8/12 | 12/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard K305 Dose (N=12) | High K305 Dose (N=12)
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Blood pressure diastolic increased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 0 | 1
Headache (Nervous system disorders) | 3 | 3
Sinus headache (Nervous system disorders) | 1 | 0
Euphoric mood (Psychiatric disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 9
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 | 9 — Runny nose
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No